CLINICAL TRIAL: NCT02398149
Title: Characterizing Upper Extremity Function in Individuals With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Mount Sinai Rehabilitation Hospital (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Jennifer Ruiz, DPT, Research Manager, Mandell MS Center, Mount Sinai Rehabilitation Hospital
Other Study IDs: 13-12-002-E; RG 4815A2/2 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2015-03-02; First posted 2015-03-25 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PwMS receiving care at the Mandell Center

SUMMARY:
Upper extremity (UE) function is critical to maintaining independence. Better understanding of UE involvement in MS will provide necessary information to prioritize the design and selection of future interventions. The goal of the proposed project is to characterize UE involvement in a population of community-based persons with MS across the International Classification of Functioning, Disability & Health (ICF) domains and constructs.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical Clinical diagnosis of MS
* Receive MS care at the Mandell MS Center
* Cognitively able to understand directions and complete protocol
* Signed consent form approved by the Saint Francis Institutional Review Board
* 18 years of age or older

Exclusion Criteria:

* Unwilling or unable to complete assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with MS who receive care at the Mandell Center for Multiple Sclerosis.
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Prevalance of Impairment in the Upper Extremity | 3hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mandell Center for Multiple Sclerosis at the Mount Sinai Rehabilitation Hospital, Hartford, Connecticut, United States